CLINICAL TRIAL: NCT03472443
Title: Sinew Acupuncture for de Quervain's Tenosynovitis: a Randomised Controlled Trial
Brief Title: Sinew Acupuncture for de Quervain's Tenosynovitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UW 18-013
Record Dates: First submitted 2018-03-05; First posted 2018-03-21 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2018-05

CONDITIONS: de Quervain's Tenosynovitis
MeSH Terms: conditions — De Quervain Disease | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sinew Acupuncture (Experimental)
  Interventions: Other: acupuncture
- Waitlist (No Intervention)

INTERVENTIONS:
Other: acupuncture — Subjects will receive Sinew Acupuncture 2-3 times in two weeks, a total of 5 sessions. Needles will be inserted into the Sinew Acupoints on the affected wrist and forearm. Needles will be inserted along the subcutaneous level, nearly parallel to the skin, and the tip of needles pointing towards the painful spot at the radial styloid. 4-6 sinew acupoints will be used.
  Arms: Sinew Acupuncture

SUMMARY:
Background:

Prevalence of de Quervain's Tenosynovitis (dQt) is estimated at 0.5% among men and 1.3% among women. As there is an increasing length of time in smart phone usage, the prevalence is believed to be higher in the future. However, the public has a common avoidance of corticosteroid usage.

Although the surgical treatment of the disease is reported to be effective in providing long term relief, its complications include radial sensory nerve injury, incomplete decompression, and volar subluxation of the tendons. The above factors raised the need of alternative treatments.

Sinew Acupuncture is a new acupuncture technique developed based on the Jing-jin theory from "Huangdi Neijing" the tradition Chinese Medicine classic literature. Previous observational studies indicated that sinew acupuncture had the immediate analgesic effect on soft tissue injuries at various locations. It is a subcutaneous and transverse needling which minimizes the pain, sore, swelling sensations of acupuncture. A controlled study includes longer follow-up is needed for providing evidence for this alternative treatment , which is safe and with the least undesired sensation.

Aims:

1. To determine whether sinew acupuncture can reduce pain (measured by Visual Analogue Scale VAS) of dQt patients.
2. To determine whether sinew acupuncture can reduce disability (measured by pinch strength, grip strength and the Quick Disabilities of the Arm, Shoulder, and Hand Q-DASH questionnaire ) of dQt patients.
3. To determine whether sinew acupuncture can improve life quality (measured WHOQOL-BREF Quality of Life Questionnaire) of dQt patients

Design:

A randomised subject trial will be employed. A total of 68 cases will be recruited in the study and allocated into study and wait-list control group under ratio 1:1. Treatment group participants will receive 5 treatments in 2 weeks and follow-up sessions after 6 and 12 weeks. Wait-list control group participants will receive same treatment and assessment after waiting and follow-up period. Both groups will receive health education session on dQt. The subjects are prohibited from receiving corticosteroid injection for treating de Quervain's Tenosynovitis. The subjects are recommended not to receive any other treatments for dQt during the trial period; Rescue medication for pain is allowed if patients have intolerant pain. Any treatments or medications for dQt received should be reported and recorded.

Setting:

The Hong Kong Tuberculosis Association - The University of Hong Kong Chinese Medicine Centre for Training and Research (Aberdeen)

Participants: 68 subjects with dQt

Treatment:

According to the theory of Sinew Acupuncture, acupoints are chosen based on 3 criteria, 1. the tender spots, 2.the spots which induce relief of symptoms and 3.the "knots" (elevated spots of the soft tissues, can be located by Chinese Medicine Practitioner (CMP) with Sinew Acupuncture training), these spots should locate along the "Jing-Jin" where the diseased spot lies, in this case the "Jing-Jin" of the Lung meridian and the Large Intestine meridian. Acupoints chosen for Sinew Acupuncture should lie within the forearm area. Subcutaneous acupuncture with the needle tips pointing towards the radial styloid activates the "Wei-Qi" to achieve analgesic effect and to promote healing.

Measures:

Primary outcome: change of Visual Analogue Scale (VAS) score in the 5th treatment (week 2) from baseline.

secondary outcome: Q-DASH (Quick Disabilities of the Arm, Shoulder, and Hand), WHOQOL-BREF Quality of Life Questionnaire, pinch strength, grip strength and averse events.

Data analysis:

The scores of VAS and Q-DASH at different time points are reported as means ± standard deviation. The scores are analysed by the intent-to-treat analysis. The last observation carried forward analyses will be employed for missing value. The difference between two groups at a time point or the difference between the two time-points in a group is tested by the student t-test. The level of the statistical significance is set P<0.05. Subgroup analysis and multiple regression analysis will be conducted to eliminate the possible bias due to the length of waiting time, the use NSAIDs, or other factor.

ELIGIBILITY:
Inclusion Criteria:

* people aged ≥18 years who have clinically diagnosed de Quervain's Tenosynovitis on one or both wrists based on the discrete tenderness of the first extensor compartment and a positive Finkelstein test.
* pain persisting for ≥3 months,
* with an average ≥40 mm in VAS in the week prior to the screening visit.

Exclusion Criteria:

* subjects who have possible traumatic or neoplastic origin of symptoms, subjects who have uncontrolled concomitant disease (such as diabetes mellitus or coagulopathy),
* prior treatment in the last 4 weeks with acupuncture, Tuina, physiotherapy, extracorporeal shock wave therapy, low-level laser therapy, steroid injection and/or surgery at the same anatomical location,
* inability to fill in follow-up forms or absence of self-determination in the participating patient.
* subjects who are pregnant.
* serious mental problem, SLUMS≤19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 2 weeks
  The horizontal VAS is a pain scale consisting of a 100-mm long horizontal line with the anchors "no pain" on the left side (0 mm) and "worst imaginable pain" on the right side (100 mm).

SECONDARY OUTCOMES:
Quick Disabilities of the Arm, Shoulder, and Hand (Q-DASH) questionnaire | up to 12 weeks
  The Q-DASH is a 11-item questionnaire to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb, scored 0 (no disability) to 100.
Pinch strength | up to 12 weeks
  Pinch strength will be assessed by a Jamar Hydraulic Pinch Gauge. The value is presented in kilogram.
Grip strength | up to 12 weeks
  Grip strength will be assessed by a Jamar dynamometer. The value is presented in kilogram.
Quality of Life Questionnaire | up to 12 weeks
  WHOQOL-BREF Quality of Life Questionnaire comprises 26 items, which measure the four domains: physical health, psychological health, social relationships, and environmental health. Each individual item of the WHOQOL-BREF is scored from 1 to 5 on a five-point likert scale. The scores are then transformed linearly to a 0-100-scale. The higher total scores denote higher quality of life.
Adverse events | 2 weeks
  Adverse events and safety issues

CONTACTS AND LOCATIONS:
Overall Officials: Haiyong Chen, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The Hong Kong Tuberculosis, Association The University of Hong Kong Clinical Centre for Teaching and Research in Chinese Medicine, Aberdeen, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Will share the data after the publication.

REFERENCES:
- [Result] Leung K, Ma OC, Qin Z, Ting H, Lau AH, Lun KK, Chan HY, Wen GY, Ng JT, Chow L, Chu CY, Ho TS, Tsang K, Ng BFL, Fok MWM, Fang CXS, Lao L, Chen H. Acupuncture for de Quervain's tenosynovitis: A randomized controlled trial. Phytomedicine. 2022 Sep;104:154254. doi: 10.1016/j.phymed.2022.154254. Epub 2022 Jun 14. PMID 35728386
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35728386/